CLINICAL TRIAL: NCT04295603
Title: Impacts of Touch-massage on the Experience of Patients With Chronic Pain and on the Provider-patient Relationship in Inpatient Settings: a Mixed Method Study.
Brief Title: Impacts of Touch-massage on the Experience of Patients With Chronic Pain: a Mixed Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Gora Da Rocha, Professor assistant, School of Health Sciences Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-00848
Record Dates: First submitted 2020-02-17; First posted 2020-03-04 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain
Keywords: Toucher-Massage; Well-being; Gratitude
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Monocentric study with a design of non-randomized cluster trial. The treatment is assigned to one of two care units and subjects are allocated to the care unit not according to a randomization process but based on administrative basis.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toucher Massage intervention (Experimental): The intervention for the Experimental Group (EG) includes a massage time of about 15 minutes on the foot area .
  Interventions: Other: Toucher Massage (TM) on the feet
- Homedics Machine intervention (Experimental): The Control Group (CG) will benefit from an intervention of identical duration. The treatment consists of a foot massage with a Homedics HM MP RELEX 90 device, a heat-free "shiatsu" program, which lasts about 15 minutes.
  Interventions: Other: Homedics HM MP RELEX 90 device

INTERVENTIONS:
Other: Toucher Massage (TM) on the feet — The intervention for the Experimental Group (EG) includes a massage time of about 15 minutes (according to current Geneva Hospital practice) on the foot area. At least four sessions will be delivered and spread over two weeks. The TM will be provided by the care team. The training time for the workers corresponds to 2 times 2 hours. In order to be as close as possible to a standardized session, practitioners will benefit from an intervention guide.
  Arms: Toucher Massage intervention
Other: Homedics HM MP RELEX 90 device — The Control Group (CG) will benefit from an intervention of identical duration. The treatment consists of a foot massage with a Homedics HM MP RELEX 90 device, a heat-free "shiatsu" program, which lasts about 15 minutes. The use of the Homedics device is no more a common treatment than the practice of Touch-Massage. TM involves a therapeutic relationship between caregiver and patient. It is for this reason that we need a comparator that should allow us to keep the aspect of the massage while decreasing the aspect of the therapeutic relationship and therefore offer us an adequate comparator.
  Arms: Homedics Machine intervention

SUMMARY:
The main purpose of this study is to evaluate the impacts of Toucher-Massage on the experience of patients with chronic pain. The study takes place in two rehabilitation internal medicine services of the University Hospitals of Geneva at 2 inpatients units with 78 participants (39 per group).

DETAILED DESCRIPTION:
This is a monocentric study with a design of non-randomized cluster trial with an exploratory qualitative part. The treatment is assigned to one of two care units and subjects are allocated to the care unit not according to a randomization process but based on administrative basis.

The main purpose of this study is to evaluate the impacts of Toucher-Massage (TM) on the experience of patients with chronic pain hospitalized in two rehabilitation internal medicine services.

The main objective is to measure the effects of TM on the global impression of change of the perception of pain.

The secondary objectives are:

1. Measure the effects on

   1. the severity and impact of pain
   2. anxiety/depression
   3. caregiver-patient interaction
2. Explore the experiences of patients benefiting from TM
3. Explore perceptions, resistance, barriers and facilitators regarding the proposed interventions with the health care teams of the units.

The population is patients suffering from chronic pain in two units of the internal medicine rehabilitation service at Beau-Séjour. The two units are similar in terms of care intake and populations cared for.

The required sample size is 78 participants (39 per group)

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for a minimum of two weeks
* Suffering from chronic pain for more than 3 months
* Having sufficient command of French in reading, writing or speaking

Exclusion Criteria:

* Documented cognitive impairments, and jeopardizing their ability to discern
* Diagnosed with cancer that does interfere with foot massage (extremities metastases)
* Dermatological conditions that interfere with foot massage
* Suffering from major polyneuropathy
* Taking anticoagulants or bleeding disorders
* Being pregnant
* Having a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Global impression of change | Baseline, two weeks
  Global impression of change will be measured by The Patient Global Impression of Change (PGIC).
  Minimum value = 1 (no change or condition has got worse) Maximum value = 7 (a great deal better, and a considerable improvement that has made all the difference)

SECONDARY OUTCOMES:
Severity of pain | Baseline, two weeks
  The Brief Pain Inventory (BPI) assesses the severity of pain and the impact on activities. The scale contains nine items: four of which have a numerical assessment scale for pain severity ranging from 0-10 (0= no pain and 10 representing the strongest possible). The impact of pain is assessed on general activity activities, mood, walking ability, work, relationships, sleep, and taste for life (0= does not interfere, 10= gene completely). The scale provides two main scores: a severity score and a pain repercussions score.
Anxiety, depression | Baseline, two weeks
  The Hospital Anxiety and Depression Scale (HADS) is composed of seven items measuring anxiety, and seven items concerning depression.
  Minimum value= 0 (never) Maximum value = 3 (really very often). A score greater than or equal to 11 indicates that the person is suffering from anxiety or depression.
The patient's perception of their interaction with the caregiver | Baseline, two weeks
  The Nurse-Patient-Interaction Scale (NPIS) questionnaire will be used to assess the patient's perception of interaction with caregivers across 14 items.
  Minimum value = 1 (not at all) Maximum value = 10 (a lot). The higher the score, the better the interaction with caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Jules Desmeules, PhD, Principal Investigator — University Hospital, Geneva; Christine Cedraschi, PhD, Principal Investigator — University Hospital, Geneva; Catherine Bollondy Pauly, MSc, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Haute Ecole de Santé, Geneva
  - Hôpitaux Universitaires de Genève, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Da Rocha Rodrigues MG, Bollondi Pauly C, Thentz C, Boegli M, Curtin F, Luthy C, Cedraschi C, Desmeules J. Impacts of Touch massage on the experience of patients with chronic pain: A protocol for a mixed method study. Complement Ther Clin Pract. 2021 May;43:101276. doi: 10.1016/j.ctcp.2020.101276. Epub 2020 Nov 28. PMID 33548750